CLINICAL TRIAL: NCT05019157
Title: TELE - WEAR: a Multi - Centre, Blinded, Randomized Controlled Trial Investigating the Efficacy, Efficiency and Cost - Effectiveness of a Cardiac Telerehabilitation Program Using Wearable Sensors (TELE - WEAR). Rationale and Study Design
Brief Title: Cardiac Telerehabilitation Effectiveness Using Wearable Sensors
Acronym: TELE-WEAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Garyfallia Pepera (Other)
Responsible Party: Sponsor-Investigator, Garyfallia Pepera, Clinical Professor, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 364/01-06-2021
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Cardiac Rehabilitation; Telerehabilitation
Keywords: wearable sensors; exercise training; functional capacity
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: supervised, randomised controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation group (Experimental): Participants will undertake the first three training sessions in the outpatient clinic under the supervision of the specialized staff for familiarization with the intervention. and then the participants will proceed with the telerehabilitation program at their homes. Participants will undergo an exercise - based program 3 times/week, comprised of 10' warm up exercises, 40' aerobic, resistance and balance exercises and 10' cool down, with the use of wearable sensors.
  Interventions: Other: Telerehabilitation group
- Centre - based rehabilitation group (Active Comparator): Participants will attend an exercise - based cardiac rehabilitation program at the outpatient clinic's facilities under the supervision of cardiac rehabilitation specialized staff. The participants will receive an individually tailored training program on a treadmill or a cycle ergometer 3 times/week, comprised of 10' warm up exercises, 40' aerobic, resistance and balance exercises and 10' cool down.
  Interventions: Other: Centre - based rehabilitation group
- Usual care group (No Intervention): Patients will not undertake any exercise based intervention and will only follow their usual medication treatment .The patients will wear the accelerometer for the 12 week study duration and visit the corresponding outpatient cardiac clinic every 4 weeks to upload the recorded data. The patients will also receive educational phone videoconference sessions every week for physical activity, diet/nutritional and smoking cessation counseling.

INTERVENTIONS:
Other: Telerehabilitation group — Participants will undertake the first three training sessions in the outpatient clinic for familiarization with the training modalities, the wearable sensors and the data uploading. Afterwards, the participants will proceed with the telerehabilitation program at their homes. The participants will be lent the wearable sensors and will undergo an exercise - based program 3 times/week, comprising of 10' warm up exercises, 40' aerobic, resistance, balance exercises and 10' cool down.Training sessions will be monitored, in real time, by the study investigator. Participants should upload the recorded data to Polar Flow web platform after every training session and should visit the outpatient clinic every month to upload the accelerometry's recorded data to a secure personal computer) application. Educational and informational videoconferences will be held every week for upright training exercise sessions, physical activity counseling, diet/nutritional and smoking cessation counseling.
  Arms: Telerehabilitation group
Other: Centre - based rehabilitation group — Participants will attend an exercise - based cardiac rehabilitation program at the outpatient clinic's facilities under the supervision of cardiac rehabilitation specialized staff. The participants will receive an individually tailored training program on a treadmill or a cycle ergometer. Total training attendance rate will be documented by the cardiac rehabilitation centre staff. Patients will be instructed to wear a tri - axial accelerometer during the entire 12 weeks study period. Participants should upload recorded data to the local server every month. Educational videoconferences will be held every week for physical activity counseling, diet/nutritional and smoking cessation counseling.
  Arms: Centre - based rehabilitation group

SUMMARY:
Objective: To evaluate the efficacy, efficiency and cost - effectiveness of a cardiac telerehabilitation program using wearable sensors

Design: Supervised single-blinded randomized controlled trial, comparing three groups, with follow-ups at baseline, 12 weeks (completion of the intervention), 6 months after the completion of the intervention

Setting: cardiac rehabilitation centres, patients home environments Participants: A total of 102 cardiac patients, regardless sex, aged 18 years and older were randomly assigned to a telerehabilitation group (n = 34), a centre - based cardiac rehabilitation group(n=34) and a usual care control group (n = 34).

Interventions: Exercise - based cardiac rehabilitation program for the intervention groups (both in cardiac clinics' settings and in patients' homes) consisted of three sessions each week for 12 consecutive weeks. The control group received no exercise intervention.

Measurements: Main outcome was measured by Cardiopulmonary Exercise Testing. Secondary outcomes were measured by accelerometry and the use of proper questionnaires.

DETAILED DESCRIPTION:
Methods Research design

A supervised, single - blind, randomized controlled trial design will be used to examine the efficacy, efficiency and cost - effectiveness of a cardiac telerehabilitation program using wearable sensors. The study was approved by the ethics committee of University of Thessaly.

Sample One hundred and two (102) cardiac patients will be recruited from cardiac rehabilitation centres. Subject eligibility criteria are: a) 18 years of age and older b) diagnosis of stable cardiovascular diseases, acute coronary syndrome, coronary artery bypass grafting within the previous six months c) ability to perform physical exercise d) ability to understand and write in the Greek language e) possession of a mobile smartphone and access to internet facilities.

Assessments Study data will be collected at baseline, the completion of the intervention period (12 weeks follow - up) and 6 months after the completion of the intervention (long - term follow - up)

Procedure

The telerehabilitation group will undergo a telemonitored exercise - based rehabilitation program 3 days a week for 12 consecutive weeks for 60'/session. The centre - based rehabilitation group will undertake a supervised exercise - based rehabilitation program 3 days a week for 12 consecutive weeks for 60'/session at the rehabilitation centres' facilities. The control group will not receive any exercise intervention during that period.

Outcome measures Functional ability, as the primary outcome of the study, will be assessed at baseline, at 12 weeks and 6 months after the completion of the intervention (long - term follow - up) via cardiopulmonary exercise testing.

Physical activity will be recorded and evaluated at the 12 weeks follow up andn the long - term follow - up by the use of tri - axial accelerometer and the International Physical Activity Questionnaire (IPAQ).

Quality of life will be assessed at baseline, at 12 weeks and 6 months after the completion of the intervention (long - term follow - up) by the use of Health related quality of life Questionnaire(HRQoL).

Anxiety levels and smoking cessation will be evaluated at baseline, at 12 weeks and 6 months after the completion of the intervention (long - term follow - up) through the use of the Hospital Anxiety and Depression scale (HADS) and the fagerstrom Test for Nicotine Dependence (FTND) respectively.

Training adherence will be evaluated during the 12 week assessment endpoint, taking in account the total number of successfully completed training sessions.

The cost-effectiveness analysis will be performed using the assessment of Quality-adjusted life years (QALYs) as a utility measure, obtained with the EuroQol-5D questionnaire at baseline and 12 - weeks follow - up assessment

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≥18 years
* stable cardiovascular disease ; acute coronary syndrome; coronary artery bypass grafting within the previous six months
* ability to perform physical exercise,
* to speak, read and write Greek
* possession of a mobile phone/smartphone
* internet access at home

Exclusion Criteria:

* ventricular arrhythmia or myocardial ischemia during low to moderate exercise intensity as assessed by symptom limited exercise testing at baseline
* heart failure New York Heart Association (NYHA) class IV
* comorbidity precluding exercise training (e.g. orthopaedic, neurological or cognitive conditions)
* acute myocardial infarction (within two days)
* stenosis
* unstable angina
* uncontrolled atrial or ventricular arrhythmia
* aortic uncontrolled congestive heart failure
* acute pulmonary embolism
* acute myocarditis or pericardial effusion
* uncontrolled diabetes mellitus (Type I, II)
* hemodynamic instability or exercise-induced arrhythmia in baseline (initial) assessment
* severe obstructive respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in the levels of physical fitness | Baseline, 12 week follow - up (end of intervention), 6 months after the completion of the intervention
  Physical fitness will be assessed in all study groups by peak oxygen uptake, determined by cardiopulmonary exercise testing (CPET) with respiratory gas analysis at the outpatient clinic.

SECONDARY OUTCOMES:
Change in the levels of physical activity | 12 week follow - up (end of intervention), 6 months after the completion of the intervention
  Daily physical activity (PA) is defined as the total number of daily low - intensity and high - intensity steps as measured objectively from a tri-axial accelerometer and subjectively through the use of the International Physical Activity Questionnaire.
Change in the Quality of participants' lives | Baseline, 12 week follow - up (end of intervention), 6 months after the completion of the intervention
  Assessment of the participants' quality of life will be evaluated with the use of the Health Related Quality of Life questionnaire (HRQoL).
Cost - effectiveness | 12 week follow up
  The cost-effectiveness analysis will be performed using the assessment of Quality-adjusted life years (QALYs) as a utility measure. Patients will complete the European Quality of Life Five Dimension (EuroQol-5D) individually and their final scores will be converted into QALYs. The cost / benefit analysis will result from the calculation of the incremental cost-effectiveness ratio (ICER):
  ICER = (cost intervention group - cost control group) / (effectiveness intervention group - effectiveness control group).
  Incremental cost refers to the difference, per patient, in the total average cost between the intervention groups and the control group. Incremental effectiveness was defined as the difference in the mean change in QALYs between the intervention group and the control group.
Adherence to rehabilitation program | 12 week follow up
  Patients' training adherence is defined as a percentage counted from the total number of completed training sessions. Patients' adherence in the telerehabilitation group will be evaluated through the Polar Flow web application as the overall completion rate of prescribed exercise sessions. Adherence in the centre - based cardiac rehabilitation group is determined as the number of attended training sessions at the outpatient clinic facilities, as recorded by the outpatient clinic's staff.
Change in the levels of anxiety and depression | Baseline, 12 week follow - up (end of intervention), 6 months after the completion of the intervention
  Anxiety and depression rates will be assessed through the Hospital Anxiety and Depression Scale (HADS) which has seven items for the depression subscale and seven items for the anxiety subscale. Scoring for each item ranges from zero(0) to three(3), with three(3) denoting highest anxiety or depression/anxiety level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Change in the smoking behaviour | Baseline, 12 week follow - up (end of intervention), 6 months after the completion of the intervention
  Smoking cessation will be evaluated through the use of the fagerstrom Test for Nicotine Dependence(FTND).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antoniou V, Xanthopoulos A, Giamouzis G, Davos C, Batalik L, Stavrou V, Gourgoulianis KI, Kapreli E, Skoularigis J, Pepera G. Efficacy, efficiency and safety of a cardiac telerehabilitation programme using wearable sensors in patients with coronary heart disease: the TELEWEAR-CR study protocol. BMJ Open. 2022 Jun 23;12(6):e059945. doi: 10.1136/bmjopen-2021-059945. PMID 35738643